CLINICAL TRIAL: NCT05259995
Title: Verification of Performance of Sustained Acoustic Medicine Device Designs Diathermy
Brief Title: Sustained Acoustic Medicine Ultrasound Diathermy Clinical Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DT-01-2022
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Measurement of Diathermy on Anatomical Locations of the Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sustained Acoustic Medicine Device Group 1 (Experimental): Patients receive treatment from the SAM Ultrasonic Diathermy Device 1 for 4 hours. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Medicine
- Sustained Acoustic Medicine Device Group 2 (Active Comparator): Patients receive treatment from the SAM Ultrasonic Diathermy Device 2 for 4 hours. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Medicine

INTERVENTIONS:
Device: Sustained Acoustic Medicine — The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity delivering 18,720 Joules of ultrasound per 4 hour treatment.
  Other Names: SAM; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device; Long Duration Low-Intensity Device

SUMMARY:
The purpose of this study is to measure diathermy performance of Sustained Acoustic Medicine Devices with commercially available ultrasound gel coupling patches.

ELIGIBILITY:
Inclusion Criteria:

• Healthy Volunteer

Exclusion Criteria:

* Is pregnant/nursing.
* Has an active infection, open sores, or wounds in the treatment area.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Ultrasound Diathermy (Degrees Centigrade) | 0 - 4 hours
  Temperature Measurement On Body (Degrees Centigrade)

CONTACTS AND LOCATIONS:
Overall Officials: George Lewis, PHD, Principal Investigator — ZetrOZ, Inc.
Locations (1):
- ZetrOZ, Trumbull, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigby JH, Taggart RM, Stratton KL, Lewis GK Jr, Draper DO. Intramuscular Heating Characteristics of Multihour Low-Intensity Therapeutic Ultrasound. J Athl Train. 2015 Nov;50(11):1158-64. doi: 10.4085/1062-6050-50.11.03. Epub 2015 Oct 28. PMID 26509683